CLINICAL TRIAL: NCT05136339
Title: Healthy Immigrant Community: Mobilizing the Power of Social Networks
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Mark L Wieland, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 21-009339; P50MD017342-01 (NIH)
Record Dates: First submitted 2021-11-16; First posted 2021-11-29 (Actual); Results first posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Weight Loss
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Community-Based Mentoring and Education Sessions (Experimental): Subjects will receive the intervention of community-based mentoring and education sessions immediately after enrollment.
  Interventions: Behavioral: Community-based mentoring and education sessions
- Delayed Community-Based Mentoring and Education Sessions (Experimental): Subjects will receive the intervention of community-based mentoring and education sessions approximately 12 months after enrollment.
  Interventions: Behavioral: Community-based mentoring and education sessions

INTERVENTIONS:
Behavioral: Community-based mentoring and education sessions — Community-based mentoring and education sessions, group activities, and application of a community toolkit for healthy weight loss delivered by trained Health Promoters from Hispanic and Somali communities to their social networks.

SUMMARY:
The objective of this study is to leverage existing social networks for health behavior change relevant to obesity and cardiovascular risk among immigrant populations in Southeast, Minnesota.

ELIGIBILITY:
Inclusion Criteria:

* Self-identification as Hispanic or Somali.
* Member of a social network identified in the social network analysis.
* Willingness to participate in all aspects of the study.
* Provision of informed consent.

Exclusion Criteria:

* Pregnancy at the time of enrollment.
* Serious medical conditions or disabilities that would make physical activity difficult.
* To avoid stigmatization, a normal weight (BMI<25) will not exclude individuals from participating in the intervention, but they will be excluded from the measurements and analyses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 475 (Actual)
Dates: Start 2022-04-23 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Wieland, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Tranby B, Sia I, Clark M, Novotny P, Lohr A, Suarez Pardo L, Patten C, Iteghete S, Zeratsky K, Rieck T, Molina L, Porraz Capetillo G, Ahmed Y, Dirie H, Wieland M. Self-Efficacy Is Associated with Health Behaviors Related To Obesity and Cardiovascular Risk Among Hispanic/Latinx and Somali Immigrants To the United States. J Immigr Minor Health. 2025 Dec 11. doi: 10.1007/s10903-025-01812-9. Online ahead of print. PMID 41379348
- [Derived] Tranby B, Sia I, Clark M, Novotny P, Lohr A, Pardo LS, Patten C, Iteghete S, Zeratsky K, Rieck T, Molina L, Capetillo GP, Ahmed Y, Dirie H, Wieland M. Self-Efficacy is Associated with Health Behaviors Related to Obesity and Cardiovascular Risk among Hispanic/Latinx and Somali Immigrants to the United States. Res Sq [Preprint]. 2025 Feb 19:rs.3.rs-6001516. doi: 10.21203/rs.3.rs-6001516/v1. PMID 40034444
- [Derived] Tranby BN, Sia IG, Clark MM, Novotny PJ, Lohr AM, Pardo LS, Patten CA, Iteghete SO, Zeratsky KA, Rieck TM, Molina L, Capetillo GP, Ahmed Y, Dirie H, Wieland ML. Negative mood is associated with sociobehavioral factors contributing to cardiovascular risk in an immigrant population. BMC Public Health. 2024 Jul 16;24(1):1911. doi: 10.1186/s12889-024-19402-z. PMID 39014369
- [Derived] Lohr AM, Pratt R, Dirie H, Ahmed Y, Elmi H, Nur O, Osman A, Novotny P, Mohamed AA, Griffin JM, Sia IG, Wieland ML. The Association Between Perceived Discrimination, Age and Proportion of Lifetime in the United States Among Somali Immigrants: A Cross-Sectional Analysis. J Immigr Minor Health. 2024 Aug;26(4):689-698. doi: 10.1007/s10903-024-01589-3. Epub 2024 Jul 18. PMID 38578534
- [Derived] Tranby BN, Sia IG, Clark MM, Novotny PJ, Lohr AM, Pardo LS, Patten CA, Iteghete SO, Zeratsky KA, Rieck TM, Molina L, Capetillo GP, Ahmed Y, Drie H, Wieland ML. Negative Mood is Associated with Sociobehavioral Factors Contributing to Cardiovascular Risk in an Immigrant Population. Res Sq [Preprint]. 2024 Mar 12:rs.3.rs-3934645. doi: 10.21203/rs.3.rs-3934645/v1. PMID 38559259
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The social networks (units of randomization) were defined as the Health Promoter (HP) and their friend/family social network members. At 0-5 months, this included 29 Hispanic and 22 Somali social networks. At 6-11 months, this included 23 Hispanic and 22 Somali social networks. At 12-24 months, this included 23 Hispanic and 22 Somali social networks.
Pre-assignment Details: The units of randomization were social networks defined by a Health Promoter and their network members. Randomization occurred after all participants were enrolled and baseline measures completed. Constrained randomization was used with the assignment selected from a set of allocations balanced on ethnicity, age, network size, and sex of the HPs.
  The period titles are referring to the time after starting intervention.
Groups:
- Immediate Community-Based Mentoring and Education Sessions: Subjects received the intervention of community-based mentoring and education sessions immediately after enrollment.
  In the first 6 months (months 0-5) health promoters facilitated 12 face-to-face or virtual group visits. Each visit targeted a specific health promotion behavior for weight loss and/or reduction of cardiovascular risk. Each group session included goal setting, review of food and/or activity tracking, and positive reflections. Strategies for weight loss included regular weigh-ins, completion of food and physical activity records, reducing portion sizes, planning meals, use of MyPlate for dietary proportions, removing problem foods from the home, increasing physical activity level, and reducing sedentary behavior. HPs supported and monitored progress of their group via six evidence-based strategies: tracking, goal setting, mindfulness, social support, problem solving, and motivation.
  Over the subsequent 6 months (months 6-11), health promoters facilitated an additional 12 virtual or face-to-face weight maintenance sessions to focus on goal setting, social support, motivation for lifestyle changes, review of food and/or activity tracking, and reflections. No new education material was provided.
- Delayed Community-Based Mentoring and Education Sessions: Subjects will receive the intervention of community-based mentoring and education sessions approximately 12 months after enrollment.
  In the first 6 months (months 12-17 from baseline) health promoters facilitated 12 face-to-face or virtual group visits. Each visit targeted a specific health promotion behavior for weight loss and/or reduction of cardiovascular risk. Each group session included goal setting, review of food and/or activity tracking, and positive reflections. Strategies for weight loss included regular weigh-ins, completion of food and physical activity records, reducing portion sizes, planning meals, use of MyPlate for dietary proportions, removing problem foods from the home, increasing physical activity level, and reducing sedentary behavior. HPs supported and monitored progress of their group via six evidence-based strategies: tracking, goal setting, mindfulness, social support, problem solving, and motivation.
  Over the subsequent 6 months (months 18-24 from baseline), health promoters facilitated an additional 12 virtual or face-to-face weight maintenance sessions to focus on goal setting, social support, motivation for lifestyle changes, review of food and/or activity tracking, and reflections. No new education material was provided.
Period: 0-5 Months
Arm/Group | Immediate Community-Based Mentoring and Education Sessions | Delayed Community-Based Mentoring and Education Sessions
Started | 246 | 229
Hispanic HP | 15 | 14
Somali HP | 11 | 11
Hispanic Participants | 131 | 115
Somali Participants | 89 | 89
Completed | 213 | 208
Not Completed | 33 | 21
Period: 6-11 Months
Arm/Group | Immediate Community-Based Mentoring and Education Sessions | Delayed Community-Based Mentoring and Education Sessions
Started | 213 | 208
Hispanic HP | 14 | 9
Somali HP | 11 | 11
Hispanic Participants | 118 | 110
Somali Participants | 70 | 78
Completed | 213 | 193
Not Completed | 0 | 15
Period: 12-24 Months
Arm/Group | Immediate Community-Based Mentoring and Education Sessions | Delayed Community-Based Mentoring and Education Sessions
Started | 213 | 193
Hispanic HP | 14 | 9
Somali HP | 11 | 11
Hispanic Participants | 116 | 103
Somali Participants | 72 | 70
Completed | 195 | 180
Not Completed | 18 | 13

BASELINE CHARACTERISTICS:
Population: The health promoters are enrolled participants and included in the baseline characteristic data.
Groups:
- Total: Total of all reporting groups
Arm/Group | Immediate Community-Based Mentoring and Education Sessions | Delayed Community-Based Mentoring and Education Sessions | Total
Number analyzed (Participants) | 246 | 229 | 475
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.9 (14.2) | 45.4 (14.2) | 45.1 (14.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 139 | 134 | 273
  Male | 93 | 87 | 180
  Other | 11 | 6 | 17
  Missing | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 146 | 129 | 275
  Not Hispanic or Latino | 99 | 98 | 197
  Unknown or Not Reported | 1 | 2 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 96 | 97 | 193
  White | 146 | 129 | 275
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 3 | 7
Region of Enrollment [Number; unit: participants]
  United States | 246 | 229 | 475
Life's Simple 6 Composite [Mean (Standard Deviation); unit: units on a scale] | 6.4 (1.9) | 6.5 (1.9) | 6.4 (1.9)
Waist Circumference [Mean (Standard Deviation); unit: Centimeters] | 101.7 (14.7) | 101.8 (12.9) | 101.7 (13.8)

OUTCOME MEASURES:

1. Primary Outcome: Change in Weight
Description: Difference in weight (measured in kilograms) from baseline to 6 months and from baseline to 12 months
Time Frame: Baseline, 6 months, 12 months
Population: The health promoters are enrolled participants and included in this outcome measure.
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Immediate Community-Based Mentoring and Education Sessions | Delayed Community-Based Mentoring and Education Sessions
Number analyzed (Participants) | 246 | 229
Kilograms
  6 months | -0.7 (9.2) | -0.4 (2.9)
  12 months | -0.7 (9.3) | -0.3 (3.7)

2. Primary Outcome: Change in Waist Circumference From Baseline to 6 Months and From Baseline to 12 Months
Description: Measured to the nearest 0.1 cm at the narrowest part of the torso between the ribs and the iliac crest.
Time Frame: Baseline, 6 months, 12 months
Population: The health promoters are enrolled participants and included in this outcome measure.
Measure: Mean (Standard Deviation); unit: Centimeters
Arm/Group | Immediate Community-Based Mentoring and Education Sessions | Delayed Community-Based Mentoring and Education Sessions
Number analyzed (Participants) | 246 | 229
Centimeters
  6 months | -0.4 (7.7) | 0.3 (6.3)
  12 months | -0.3 (8.5) | 0.5 (7.2)

3. Primary Outcome: Change in "Life's Simple 6" Composite Score From Baseline to 6 Months and From Baseline to 12 Months
Description: Adapted from the American Heart Association standards based on health assessment data. Point values are assigned to each component: 2 points for ideal, 1 point for intermediate, 0 points for poor. The total sum allows for a continuous measure of cardiovascular health ranging from poor to ideal (0-12 points).
Time Frame: Baseline, 6 months, 12 months
Population: The health promoters are enrolled participants and included in this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate Community-Based Mentoring and Education Sessions | Delayed Community-Based Mentoring and Education Sessions
Number analyzed (Participants) | 246 | 229
units on a scale
  6 months | 0.4 (1.8) | -0.1 (1.7)
  12 months | 0.5 (2) | 0.2 (1.7)

4. Primary Outcome: Lost >5% of Body Weight
Description: Number of participants in each arm who lost a clinically significant amount of weight (>5%).
Time Frame: 6 months, 12 months
Population: The health promoters are enrolled participants and included in this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Community-Based Mentoring and Education Sessions | Delayed Community-Based Mentoring and Education Sessions
Number analyzed (Participants) | 246 | 229
Participants
  6 months | 24 | 12
  12 months | 37 | 18

5. Secondary Outcome: Change in Systolic Blood Pressure
Description: Measured three times and the average of the second and third readings will be used in analyses, reported in mmHg. Change from baseline to 6 months and from baseline to 12 months.
Time Frame: Baseline, 6 months, 12 months
Population: The health promoters are enrolled participants and included in this outcome measure.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Immediate Community-Based Mentoring and Education Sessions | Delayed Community-Based Mentoring and Education Sessions
Number analyzed (Participants) | 246 | 229
mmHg
  6 months | 3 (13.5) | -0.3 (14.5)
  12 months | -0.5 (13.6) | -2.4 (13.4)

6. Secondary Outcome: Change in Fasting Glucose Level
Description: 6 hours fasting glucose blood serum level, reported in mg/dL. Baseline to 6 months and baseline to 12 months.
Time Frame: Baseline, 6 months, 12 months
Population: The health promoters are enrolled participants and included in this outcome measure.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Immediate Community-Based Mentoring and Education Sessions | Delayed Community-Based Mentoring and Education Sessions
Number analyzed (Participants) | 246 | 229
mg/dL
  6 months | 2.3 (38.1) | -2.6 (36)
  12 months | -0.1 (40.1) | -4.4 (31.8)

7. Secondary Outcome: Change in Low-density Lipoprotein (LDL)
Description: Change in LDL cholesterol blood serum level, reported in mg/dL. Baseline to 6 months and baseline to 12 months
Time Frame: Baseline, 6 months, 12 months
Population: The health promoters are enrolled participants and included in this outcome measure.
Measure: Mean (Standard Deviation); unit: mg/Dl
Arm/Group | Immediate Community-Based Mentoring and Education Sessions | Delayed Community-Based Mentoring and Education Sessions
Number analyzed (Participants) | 246 | 229
mg/Dl
  6 months | 4.9 (26.3) | 3.1 (30.8)
  12 months | -2.9 (25.3) | -1 (32.3)

8. Secondary Outcome: Change in Dietary Quality
Description: 24-hour dietary recall collected using the Nutrition Data System for Research (NDSR) used to calculate the Healthy Eating index (HEI-2015). The HEI range is 0-100 with higher scores indicating healthier dietary quality. Scores can be further categorized as HEI≥69.3 optimal, HEI 56.9-69.2 intermediate, HEI<56.9 poor. Change from baseline to 6 months and baseline to 12 months.
Time Frame: Baseline, 6 months, 12 months
Population: The health promoters are enrolled participants and included in this outcome measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Immediate Community-Based Mentoring and Education Sessions | Delayed Community-Based Mentoring and Education Sessions
Number analyzed (Participants) | 246 | 229
units on a scale
  6 months | 2.3 (18.3) | 2.3 (16.6)
  12 months | 0 (16.9) | 3.6 (17)

9. Secondary Outcome: Change in Physical Activity
Description: Measured using the International Physical Activity Questionnaire (IPAQ) that assesses the number of minutes of mild, moderate, and vigorous physical activity over the previous 7 days, scores categorized as ≥150 min/wk moderate or ≥75 min/wk vigorous or ≥150 min/wk moderate+vigorous = optimal; 1-149 min/wk moderate or 1-74 min/wk vigorous or 1-149 min/wk moderate+vigorous = intermediate; no physical activity = poor. Baseline to 6 months and baseline to 12 months. For this study, we present IPAQ results as a continuous variable of MET minutes per week, which refers to the total amount of physical activity measured in Metabolic Equivalent of Task (MET) units over a week. Physical Activity Guidelines recommend achieving 500 to 1,000 MET minutes per week for significant health benefits.
Time Frame: Baseline, 6 months, 12 months
Population: The health promoters are enrolled participants and included in this outcome measure.
Measure: Mean (Standard Deviation); unit: MET minutes per week
Arm/Group | Immediate Community-Based Mentoring and Education Sessions | Delayed Community-Based Mentoring and Education Sessions
Number analyzed (Participants) | 246 | 229
MET minutes per week
  6 months | 738.5 (3780.4) | 312.2 (4334.6)
  12 months | 290.1 (4102.2) | 1080.5 (5623.7)

10. Secondary Outcome: Change in Diastolic Blood Pressure
Description: Chage from baseline to 6 months and from baseline to 12 months (mmHg)
Time Frame: Baseline, 6 months, 12 months
Population: The health promoters are enrolled participants and included in this outcome measure.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Immediate Community-Based Mentoring and Education Sessions | Delayed Community-Based Mentoring and Education Sessions
Number analyzed (Participants) | 246 | 229
mmHg
  6 months | 0.4 (8.9) | -0.8 (9.1)
  12 months | -0.7 (8.8) | -1.9 (9.6)

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Immediate Community-Based Mentoring and Education Sessions | Delayed Community-Based Mentoring and Education Sessions
All-Cause Mortality (participants affected / at risk) | 0/246 | 0/229
Serious Adverse Events (participants affected / at risk) | 0/246 | 0/229
Other Adverse Events (participants affected / at risk) | 0/246 | 0/229

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-09-28): https://cdn.clinicaltrials.gov/large-docs/39/NCT05136339/Prot_SAP_001.pdf
  • Informed Consent Form (2021-10-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT05136339/ICF_000.pdf